CLINICAL TRIAL: NCT03657589
Title: Sonographic Imaging of Oral and Dental Anatomical Structures (A Pilot Study)
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: MICHR Pilot grant (UL1TR000433) (Unknown); Delta Dental Foundation (Other); POM Supplemental Grant (Unknown); SOD Collision Award (Unknown); AAP's SUNSTAR Innovation Grant (Other)
Responsible Party: Principal Investigator, Hsun-Liang Chan, Clinical Assistant Professor, University of Michigan
Other Study IDs: HUM00099062
Record Dates: First submitted 2018-08-30; First posted 2018-09-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Ultrasound; Oral Mucosa; Gingival Recession; Alveolar Bone Loss
MeSH Terms: conditions — Gingival Recession; Alveolar Bone Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with 1 missing tooth: Patients with 1 missing anterior or premolar tooth and planned for implant surgery were recruited. Gingiva and alveolar bone were ultrasound scanned and compared to CT scans and direct measures during implant surgery.

SUMMARY:
The overall purpose of this study is to establish an ultrasound technique to aid in oral and dental examination of soft and hard tissues. Ultrasound is currently not used in Dentistry and associated oral examinations and its usefulness for clinical practice will be explored. This study will investigate the use of ultrasonic imaging for planning and placing dental implants, as well as evaluate the use of ultrasonic imaging for monitoring marginal bone loss around dental implants.

DETAILED DESCRIPTION:
This study will involve two different groups of subjects: Patients scheduled for a dental implant procedure, and patients scheduled for a revision surgery after developing infection after implant surgery.

Twenty subjects examining only specific aim one is funded and will be studied. If future funding is granted and additional 30 subjects for aim one and 40 for aim two will be studied Subjects in both groups will receive an ultrasound examination of the oral cavity prior to their clinically-scheduled dental surgery. Subjects in group 1 also may receive a CBCT scan if not previously clinically-ordered.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years of age and older who will be scheduled to have an implant surgery from premolar to premolar with bilateral adjacent teeth present will be recruited.

Exclusion Criteria:

* Patients under 18 years of age.
* Unwilling or unable to read and sign this informed consent document.
* Do not have a tooth on each side of the implant that will be placed.
* Women who are pregnant or unsure of their pregnancy status.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects 18 years of age and older who will be scheduled to have an implant surgery from premolar to premolar with bilateral adjacent teeth present will be recruited.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-01-16 (Actual)

PRIMARY OUTCOMES:
ultrasound soft tissue thickness | At least 6 months after implant crown placement (1 time point)
  soft tissue thickness at the missing tooth gap and adjacent teeth were measured with ultrasound

SECONDARY OUTCOMES:
ultrasound alveolar bone height | At least 6 months after implant crown placement (1 time point)
  alveolar bone height at the missing tooth gap and adjacent teeth was measured

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhaskar V, Chan HL, MacEachern M, Kripfgans OD. Updates on ultrasound research in implant dentistry: a systematic review of potential clinical indications. Dentomaxillofac Radiol. 2018 Jul;47(6):20180076. doi: 10.1259/dmfr.20180076. Epub 2018 Jun 6. PMID 29791198
- [Background] Chan HL, Sinjab K, Li J, Chen Z, Wang HL, Kripfgans OD. Ultrasonography for noninvasive and real-time evaluation of peri-implant tissue dimensions. J Clin Periodontol. 2018 Aug;45(8):986-995. doi: 10.1111/jcpe.12918. Epub 2018 Jun 25. PMID 29757464
- [Background] Chan HL, Sinjab K, Chung MP, Chiang YC, Wang HL, Giannobile WV, Kripfgans OD. Non-invasive evaluation of facial crestal bone with ultrasonography. PLoS One. 2017 Feb 8;12(2):e0171237. doi: 10.1371/journal.pone.0171237. eCollection 2017. PMID 28178323
- [Background] Chung MP, Wang IC, Chan HL, Wang HL. Evaluation of Buccal Bone Concavity in the Esthetic Zone: A Cadaver Study. Implant Dent. 2017 Oct;26(5):751-755. doi: 10.1097/ID.0000000000000661. PMID 28914631
- [Background] Fu JH, Yeh CY, Chan HL, Tatarakis N, Leong DJ, Wang HL. Tissue biotype and its relation to the underlying bone morphology. J Periodontol. 2010 Apr;81(4):569-74. doi: 10.1902/jop.2009.090591. PMID 20367099